CLINICAL TRIAL: NCT05043168
Title: Kidney Histopathological Features in Patients After COVID-19 and SARS-CoV-2 Vaccination
Brief Title: Kidney Histopathology After COVID-19 and SARS-CoV-2 Vaccination
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-100682-BO-ff
Record Dates: First submitted 2021-09-10; First posted 2021-09-14 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Vaccination Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Kidney biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID-19: Polymerase Chain Reaction-positive SARS-CoV-2 infection
- Patients post-SARS-CoV-2 vaccination: Onset of kidney disease potentially relatable to SARS-CoV-2 vaccination based on clinical grounds

SUMMARY:
The study aims to summarize kidney histopathological findings in patients with coronavirus disease 2019 (COVID-19) and post-severe acute respiratory syndrome-coronavirus-type 2 (SARS-CoV-2) vaccination.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic has had substantial global morbidity and mortality. While COVID-19 is most commonly characterized as a respiratory illness, extrapulmonary manifestations are a prominent part its clinical spectrum. Kidney disease is a common finding in COVID-19, and has also been rarely described after SARS-CoV-2 vaccination. The main objective of this study is to summarize kidney histopathological findings in patients with COVID-19 and post-SARS-COV-2 vaccination, in whom native kidney biopsy was performed and samples were obtained by the Nephropathology Section, Institute of Pathology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with COVID-19 when kidney biopsy was performed
* history of recent homologous or heterogenous vaccine regimen comprising either vector-based vaccines or messenger ribonucleic acid-based vaccines

Exclusion Criteria:

* Patient refuses participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary inpatient and outpatient care
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Frequency of histopathologically confirmed glomerular and tubulointerstitial diseases | Kidney biopsy obtained during COVID-19 disease and up to 3 months after SARS-CoV-2 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Wiech, MD, Principal Investigator — Nephropathology Section, Institute of Pathology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puelles VG, Lutgehetmann M, Lindenmeyer MT, Sperhake JP, Wong MN, Allweiss L, Chilla S, Heinemann A, Wanner N, Liu S, Braun F, Lu S, Pfefferle S, Schroder AS, Edler C, Gross O, Glatzel M, Wichmann D, Wiech T, Kluge S, Pueschel K, Aepfelbacher M, Huber TB. Multiorgan and Renal Tropism of SARS-CoV-2. N Engl J Med. 2020 Aug 6;383(6):590-592. doi: 10.1056/NEJMc2011400. Epub 2020 May 13. No abstract available. PMID 32402155
- [Background] Sharma P, Uppal NN, Wanchoo R, Shah HH, Yang Y, Parikh R, Khanin Y, Madireddy V, Larsen CP, Jhaveri KD, Bijol V; Northwell Nephrology COVID-19 Research Consortium. COVID-19-Associated Kidney Injury: A Case Series of Kidney Biopsy Findings. J Am Soc Nephrol. 2020 Sep;31(9):1948-1958. doi: 10.1681/ASN.2020050699. Epub 2020 Jul 13. PMID 32660970
- [Background] Bomback AS, Kudose S, D'Agati VD. De Novo and Relapsing Glomerular Diseases After COVID-19 Vaccination: What Do We Know So Far? Am J Kidney Dis. 2021 Oct;78(4):477-480. doi: 10.1053/j.ajkd.2021.06.004. Epub 2021 Jun 25. No abstract available. PMID 34182049
- [Derived] de Las Mercedes Noriega M, Husain-Syed F, Wulf S, Csala B, Krebs CF, Jabs WJ, Zipfel PF, Grone HJ, Wiech T; CoV-Kidney Investigators. Kidney Biopsy Findings in Patients with SARS-CoV-2 Infection or After COVID-19 Vaccination. Clin J Am Soc Nephrol. 2023 May 1;18(5):613-625. doi: 10.2215/CJN.0000000000000106. Epub 2023 Feb 1. PMID 36723286